CLINICAL TRIAL: NCT02745054
Title: Safety of Oral Anticoagulants Registry (SOAR): A National, Hospital-Based, Sentinel Surveillance Study of the Clinical and Economic Impact of Bleeding and Bleeding Concerns Due to the Use of Oral Anticoagulants
Brief Title: Safety of Oral Anticoagulants Registry
Acronym: SOAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Quality Foundation (Other)
Collaborators: Boehringer Ingelheim (Industry); Daiichi Sankyo (Industry); CSL Behring (Industry); Janssen Scientific Affairs, LLC (Industry); Portola Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: HQF-2016-SOAR-1
Record Dates: First submitted 2016-04-04; First posted 2016-04-20 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Blood Coagulation
Keywords: oral anticoagulants; bleeding; anticoagulation reversal
MeSH Terms: conditions — Thrombosis; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: mgt of bleeding concerns/complications of oral anticoagulants — observational study of clincians' management of patients taking oral anticoagulants and having acute significant bleeding or requiring management of bleeding risk before an emergent procedure; observation limited to index hospitalization only
  Other Names: anticoagulation emergency management; anticoagulation emergency reversal

SUMMARY:
The goal of SOAR is to characterize the clinical and economic impact of clinicians' responses to major bleeding complications and pre-procedural concerns for bleeding risk in patients treated with oral anticoagulants (warfarin, anti-Xa orals, and anti-thrombin (IIa) orals) who present to the ED or in the hospital with acute illness or injury, with the eventual aim of informing the development of improved approaches to the management of OACs in the ED.

DETAILED DESCRIPTION:
Purpose and Rationale:

Until recently, warfarin was the only oral anticoagulant (OAC) available in the US, and a substantial infrastructure has developed around its management. Over the past five years, four non-Vitamin-K antagonist oral anticoagulants (NOAC) have been approved by the FDA. The NOACs are associated with generally fewer and less severe bleeding complications, and shorter half-lives, often making management of bleeding that complicates the use of these agents less problematic than similar episodes associated with warfarin. Bleeding during NOAC therapy does occur, and patients taking NOACs sometimes require procedures that cannot be delayed, for which good hemostasis is desirable, and therefore the NOAC may delay or complicate care. The challenge of this latter issue is compounded by the lack of readily available, rapid-turnaround quantitative assays for measuring the magnitude of anticoagulation effect associated with NOAC use. From a safety perspective, the large warfarin infrastructure does not translate into useful support for use of the new NOACs; their anticoagulation impact cannot be readily monitored by simple, quick tests.

In October 2015 the first specific reversal agent for a NOAC was approved, but it is useful only for dabigatran; at present, there is no specific reversal agent for anti-Xa NOACs. Emergency care providers face many concerns and insecurities regarding the safety of warfarin and the NOACs, while working in a highly pressurized care environment, often with limited patient history and little time to consider treatment options.

Because of the unique position of the hospital ED in the US healthcare continuum, it is frequently the initial site of care for patients on OACs who develop bleeding complications. In all clinical settings, there tends to be a standardized, international normalized ratio (INR)-driven pathway for the management of warfarin-related bleeds. Many EDs and hospital pharmacies are now trying to establish similarly standardized, though not evidence-driven, pathways for NOAC-related bleeding, and eagerly await the availability of additional specific reversal agents to use in such patients.

The ED represents the key sentinel surveillance point for assessing the clinical and economic impact of bleeding concerns and complications attributable to OAC therapy. Other bleeding issues that impact the pace and nature of medical and surgical care occur in the inpatient setting, especially the ICU and surgical suite. Taken together, the hospital setting (ED plus inpatient) offers a 360-degree view of the scope, significance, and cost of OAC-related bleeds and bleeding concerns.

This registry is proposed as a large, prospective, multicenter study that identifies the clinical and economic impact of safety concerns around OAC use on evaluation and management strategies in the ED and on the inpatient units of participating hospitals. The eventual aim will be to use these data to inform the gradual development of a new, protocolized safety standard in the management of OACs in the ED.

ELIGIBILITY:
Inclusion Criteria:

1. Bleeding requiring intervention - patients must be taking an OAC and meet at least one of the following criteria:

   * Acute bleeding that is potentially life-threatening at presentation
   * Acute bleeding associated with a fall in hemoglobin level by ≥2 g/dL
   * Acute bleeding associated with a hemoglobin level of ≤8 g/dL if no baseline hemoglobin is available
   * Acute symptomatic bleeding in a critical area or organ
   * Any intracranial bleeding
   * Bleeding for which more than 8 hours of direct patient monitoring is required prior to ED disposition
   * Bleeding for which intravenous (IV) Vitamin K, fresh frozen plasma (FFP), any prothrombin complex concentrates (PCC) or activated PCC (aPCC), any specific factor replacement or reversal agent, or a parenteral hemostatic agent such as tranexamic acid is administered
   * Bleeding for which packed red blood cells (PRBCs) or platelets are transfused
2. Bleeding Concern - patients must be taking an OAC and who, without overt bleeding, meet at least one of the following criteria:

   * Diagnostic or therapeutic surgical procedure for which hemostasis is desirable (e.g., emergency laparotomy) and which, in the opinion of the treating physician, cannot be postponed at least 8 hours
   * Diagnostic or therapeutic percutaneous procedure for which hemostasis is desirable (e.g., lumbar puncture) and which, in the opinion of the treating physician, cannot be postponed at least 8 hours
   * Overdose (deliberate or accidental) of one or more OAC agents that, in the opinion of the treating physician, requires the administration of Vitamin K, FFP, any PCC or aPCC, any specific factor replacement or specific reversal agent, or a parenteral hemostatic agent such as tranexamic acid, with the desire of immediate reversal of anticoagulation
   * Bleeding concern for which, in the opinion of the treating physician, more than 8 hours of direct patient monitoring is required prior to ED disposition

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for inclusion in this registry study:

* Those who have received an investigational reversal agent for an OAC during the index event (data on these patients will be collected as part the pertinent investigational study).If during the course of SOAR enrollment an investigational reversal agent is approved, and that agent is used outside a registration study, that subject is not excluded.
* Those who have received treatment for a bleed or bleeding concern at another facility immediately prior to being transferred to the enrolling facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years and older who present to the ED or hospital with an acute illness or injury and must, in the opinion of the treating clinician, be experiencing an active anticoagulation effect due to the use of an OAC, and have either:
  1. Bleeding requiring specific intervention (see below); or
  2. Bleeding concern in a non-bleeding patient requiring a specific invasive diagnostic assessment or therapeutic intervention prompting reversal, repletion or decontamination, or a clinically significant delay in intervention due to the use of an OAC (see below).
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
DESCRIPTIVE: timing endpoints: hours after presentation before any observed intervention | index hospitalization, generally less than or equal to (LTE) 7 days
  * to include time to procedure/surgery, time to infusion of one of listed medicines (PCC, aPCC, rfVIIa, idarucizumab, tranexamic acid, andexanet alfa [once approved]), type of invasive procedure/surgery, delays in procedure/surgery, relation of interventions/procedures performed to the index event, all determined by review of the medical record
  * type of invasive procedure/surgery (diagnostic/therapeutic), as documented in the medical record
  * reason for any delay in procedure, as documented in the medical record
  * procedure attributable to index event, as documented in the medical record

SECONDARY OUTCOMES:
hospital length of stay | index hospitalization only, generally LTE 7 days
  to include length of stay (LOS) in ED, hospital, and ICU, as applicable, measured in hours or days per medical record
disposition after emergency care | index hospitalization only, generally LTE 7 days
  location as documented in medical record: discharge home, admit inpatient (non-ICU), admit ICU, admit observation status, deceased
DESCRIPTIVE: blood products utilization: # units | index hospitalization only, generally LTE 7 days
  number of units of packed red blood cells, fresh frozen plasma, and/or platelets, as documented in the medical record
DESCRIPTIVE: reversal products given (with doses and timing) | index hospitalization only, generally LTE 7 days
  as per medical record, the doses and time of administration of any concentrated coagulation factors, prothrombin complex concentrate, idarucizumab, or andexanet alfa
DESCRIPTIVE: in-hospital complications: incidence, description | index hospitalization only, generally LTE 7 days
  to be classified according to surgical/medical risk
DESCRIPTIVE: costs of treatment | index hospitalization only, generally LTE 7 days
  • to include ED and total hospital costs of blood products/components, pharmaceutical products, cost of procedures (diagnostic, interventional)

CONTACTS AND LOCATIONS:
Overall Officials: Charles V Pollack, MD, Study Chair — Hospital Quality Foundation
Locations (9):
- United States (9):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Hartford Hospital, Hartford, Connecticut
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - Washington University, St Louis, Missouri
  - Kings County Hospital, Brooklyn, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Genesis HealthCare, Zanesville, Ohio
  - Reading Hospital, West Reading, Pennsylvania

IPD SHARING:
Plan to Share IPD: No